CLINICAL TRIAL: NCT03636633
Title: The Effect of Inspiratory Muscle Training and Respiratory Physiotherapy on Pulmonary Functions, Respiratory Muscle Strength and Functional Capacity in Patients With Robotic Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Aslı İrem Dönmez, PT, Research Assistant at Faculty of Health Sciences, Acibadem University, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATADEK-2018-2/55
Record Dates: First submitted 2018-08-06; First posted 2018-08-17 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Robotic Surgical Procedures; Heart Diseases
Keywords: Robotic Heart Surgery; Inspiratory Muscle Training; Pulmonary Function Test; 6-Minute Walk Test; Respiratory Muscle Strength; Functional Capacity
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Standard respiratory physiotherapy
  Patients in this group will receive standard respiratory physiotherapy two times a day, 7 days a week for 4 weeks. During hospitalization, sessions will be performed by a respiratory physiotherapist. After discharge, other sessions will be performed at home by themselves.
  Interventions: Other: Standard respiratory physiotherapy
- Training Group (Experimental): Standard respiratory physiotherapy and inspiratory muscle train
  In addition to the standard respiratory physiotherapy program, patients in this group will receive 3 sets of inspiratory muscle training with 10 repetitions twice a day for 4 weeks. During hospitalization, sessions will be performed by a respiratory physiotherapist. After discharge, other sessions will be performed at home by themselves.
  Interventions: Other: Standard respiratory physiotherapy and inspiratory muscle training

INTERVENTIONS:
Other: Standard respiratory physiotherapy — Standard respiratory physiotherapy content; diaphragmatic breathing, pursed lip breathing, segmental breathing, incentive spirometer exercises (Triflo) and coughing techniques.
  Arms: Control Group
Other: Standard respiratory physiotherapy and inspiratory muscle training — Standard respiratory physiotherapy content; diaphragmatic breathing, pursed lip breathing, segmental breathing, incentive spirometer exercises (Triflo) and coughing techniques. Addition to that, threshold IMT device will be used for the training. Training intensity will set at 40% of the maximum inspiratory pressure.
  Arms: Training Group

SUMMARY:
During the past decade, especially with the advancement of technology, major innovations and developments have been observed in the field of surgery. Cardiac surgery is one of the important area of the surgery who renews itself day by day and adds innovations to the nature in terms of patients' comfort. One of the greatest developments in cardiac surgery in this sense is the tendency to reduce the size of the incisions with less interventional procedures. Robotic surgery is getting more and more meaningful in this area. Despite the downsizing of the surgical incisions, postoperative pulmonary complications have not completely disappeared in the robotic cardiac surgery. Major respiratory problems following traditional cardiac surgery are gas exchange problems, atelectasis, decreased coughing force and sputum retention. The effectiveness of respiratory physiotherapy applied after traditional cardiac surgery for the resolution of these complications has been proved by various investigations. Inspiratory muscle training (IMT) has been found to improve autonomic modulation in heart failure patients as well as to increase inspiratory muscle strength in applied patient populations, reduce blood pressure in hypertensive patients, and increase functional capacity in elderly individuals. Considering these benefits, when inspiratory muscle training is given to people with traditional cardiac surgery, respiratory muscle strengths, respiratory functions and functional capacities are increased compared to those not given to these patients. However, although there are complications after robotic cardiac surgery, there are no studies in the literature about respiratory physiotherapy or inspiratory muscle training. Thus, the subject of this study is the comparison of the effects of standard respiratory physiotherapy and standard respiratory physiotherapy plus inspiratory muscle training on the respiratory functions, respiratory muscle strength and functional capacity of the patients with the robotic heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Being suitable for robotic cardiac surgery,
* Being hospitalized to have a robotic heart surgery,
* No complications during surgery,
* To be extubated in intensive care unite after surgery ,
* Stable clinical condition,
* To be transferred from ICU to the hospital room on the first day after surgery.

Exclusion Criteria:

* Chronic obstructive pulmonary disease,
* Unstable angina,
* Acute decompensated heart failure,
* Acute pericarditis and myocarditis,
* Complex arrhythmia,
* Uncontrolled hypertension,
* Serious orthopedic and neurological impairment,
* Uncontrolled diabetes,
* Body Mass Index > 30.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline Forced Vital Capacity (FVC) at 4 weeks | Four weeks
Change from baseline Forced Expiratory Volume in 1 second (FEV1) at 4 weeks | Four weeks
Change from baseline Peak Expiratory Flow (PEF) at 4 weeks | Four weeks
Change from baseline maximum inspiratory pressure (MIP) at 4 weeks | Four weeks
Change from baseline maximum expiratory pressure (MEP) at 4 weeks | Four weeks
Change from baseline distance covered in six-minute walk test (6MWT) at 4 weeks | Four weeks
Change from baseline carbon monoxide diffusion capacity of the lungs (DLCO) at 4 weeks | Four weeks

SECONDARY OUTCOMES:
Fatigue Severity Scale | Four weeks
  The 9 item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Assessment type: Patient reported outcomes.The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree.The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity.
Fatigue Impact Scale | Four weeks
  The fatigue impact scale was developed to assess the symptom of fatigue as part of an underlying chronic disease or condition. Consisting of 40 items, the instrument evaluates the effect of fatigue on three domains of daily life: cognitive functioning, physical functioning, and psychosocial functioning. Respondents are asked to rate the extent to which fatigue has interfered with certain aspects of their day-to-day functioning using a scale that ranges from 0 ("no problem") to 4 ("extreme problem"). Scores are then tallied to produce an overall score with a potential maximum of 160. Subscale scores can also be calculated to give a more nuanced impression of fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem MAA University Maslak Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided